CLINICAL TRIAL: NCT02669823
Title: Optimizing Sysmex Technology as an Innovative Tool to Differentiate Between Malaria (PALUdism) and BACterial Infections in a Malaria Endemic Region
Acronym: PALUBAC
Status: Completed | Type: Observational
Sponsor: Sysmex Europe GmbH (Industry)
Collaborators: Clinical Research Unit of Nanaro (CRUN), Burkina Faso (Unknown); Instituut voor Tropische Geneeskunde (ITG), Belgium (Unknown); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: PALUBAC
Record Dates: First submitted 2016-01-26; First posted 2016-02-01 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Tropical Infectious Diseases
Keywords: Diagnosis
MeSH Terms: conditions — Disease | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Children <15y: no intervention
  Interventions: Other: None, treatment as actual best practice
- Adults >=15y: no intervention
  Interventions: Other: None, treatment as actual best practice

INTERVENTIONS:
Other: None, treatment as actual best practice

SUMMARY:
Severe malaria and bacterial Blood Stream Infections (bBSI) are impossible to differentiate clinically. This poses a particular threat in low resource areas, where bBSI is often not diagnosed due to the unavailability of rapid diagnostic means. Even if used appropriately, the sensitivity of blood culture to diagnose bBSI is estimated to be around 50%. To counter the high mortality rate associated with bBSI, antibiotics are often prescribed without microbiological confirmation. Sysmex Company has developed technology that enables the rapid diagnosis of malaria using a venous blood sample. In addition algorithms based on hematological parameters can be used to monitor disease severity and progression, as well as guide further diagnostic testing based on differences seen in these parameters between various types of disease. The algorithms have been developed and tested in adult populations from different industrialized countries and in one Asian population. However no data are available neither from pediatric patients, nor from the sub-Saharan setting where the epidemiology of infectious diseases is very different from the tested settings. The objective of the study is to: 1) Assess the sensitivity and specificity of the Sysmex hematology analyzer based on the new technology to diagnose malaria in subjects older than 3 months, who present with an acute severe febrile illness in a malaria endemic area in sub-Saharan Africa 2) Test and optimize the value of Sysmex analyzers in disease diagnosis and monitoring in children older than 5 years and adults, who present with an acute severe febrile illness in a malaria endemic region in sub-Saharan Africa, to differentiate between severe malaria and bBSI, or a combination of these infections. 3) Explore the value of Sysmex analyzers in disease diagnosis and monitoring in children between 3 months and 5 years of age, who present with an acute severe febrile illness in a malaria endemic region in sub-Saharan Africa.

DETAILED DESCRIPTION:
Analytical plan

Sysmex will be blinded to:

* All clinical data except age and gender of the participant
* All laboratory and imaging data that is not obtained by the XN-analyzers.

The clinical study team will be blinded to:

- Data from the XN-analyzers, excepting the currently validated data that is used for routine patient care (e.g. total blood count, white blood differentiation)

Two researchers from Sysmex and two researchers from the study team will use the data available to them (i.e. the data to which they are not blinded) to categorize each patient according to the following categories (independently from each other) using the predefined case definitions as mentioned above.

1. Confirmed malaria parasitemia
2. Confirmed bacterial infection
3. Confirmed viral infection
4. Suspected malaria
5. Suspected bacterial infection
6. Suspected viral infection
7. Mixed infection (specified which combination)
8. No infection

Analysis for primary outcome measures

1. Diagnostic sensitivity and specificity of blue laser compared to microscopy/PCR
2. ROC curve to assess best cut-off for the blue laser based on clinical samples
3. Linear regression analysis to compare quantification of parasitemia by blue laser to microscopy/PCR
4. Compare performance of the blue laser to performance of RDT (in comparison to microscopy/PCR)
5. Diagnostic sensitivity and specificity of infection manager to detect bBSI in participants of 5 years and older.
6. Diagnostic sensitivity and specificity of the infection manager to detect bBSI combined with malaria in participants of 5 years and older.

Case definitions:

Malaria parasitemia is defined as the presence of one or more parasites in malaria microscopy or a malaria qPCR 18S result over 50 p/ml

Bacterial bloodstream infection is defined as growth of a clinically significant bacterial organism from blood culture within 5 days of incubation or a (16s) PCR result positive for a clinically significant organism

Lower respiratory tract infection: a clinical suspicion including cough and/or shortness of breath, supported by results from chest exam and chest X-ray.

Abscess: in case of superficial abscesses clinical presentation must be confirmed by pus upon drainage. In case of deep abscesses the clinical presentation must be confirmed by echography.

Meningitis: A clinical suspicion with decreased conscience and neck stiffness, confirmed by culture or agglutination performed on cerebrospinal fluid.

Pelvic inflammatory infection: Typical clinical presentation with vaginal discharge

Protrude skin infections: clinical presentation combined with a grown pathogen in skin culture or presence of pus.

Bacterial gastro-enteritis: Patients with diarrhoea and a grown pathogen from stool culture.

Urinary tract infections: Patients clinical signs of a urinary tract infection and a grown pathogen from urine culture.

Obvious causes of fever include superficial skin infection, superficial abscesses, otitis, pharyngitis and tonsillitis.

Viral infections will be diagnosed based on clinical suspicion and confirmed using PCR or serology.

ELIGIBILITY:
Inclusion Criteria:

1. Children between ages >3 months and < 15 years old OR adults of 15 years and above
2. AND willing and able to provide written informed consent (parent's or guardian's consent for minors). In case of very sick adults not able to give consent, sampling will be done and ICF will be asked upon his/her recovery or from his/her representative in case of death.
3. AND presenting with one of the following:

   Recorded temperature of > 38.0°C or temperature < 35.5°C (tympanic). OR episode of fever within 48 hours prior to admission

   OR signs of severe clinical illness including one or more of the following:
   * Respiratory distress
   * Prostration
   * Altered consciousness
   * Convulsions (one or more episodes)
   * Clinical jaundice
   * Signs of shock
   * Severe malnutrition with severe anemia (hemoglobin < 5 g/dl)
4. AND Having one of the following clinically suspected infections

   * Severe malaria
   * Invasive bacterial infection (including pneumonia, arthritis, peritonitis, meningitis or complicated urinary tract infection, typhoid fever)
   * Severe viral infection such as influenza

Exclusion Criteria:

• Fever episode for more than 7 days or no informed consent was given

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting at the district health center with suspicion of infectious disease. Since the amendment which passed in November 2016 this includes outpatients as well as inpatients.
Sampling Method: Non-Probability Sample
Enrollment: 930 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
• Diagnostic sensitivity and specificity of Sysmex XN blue laser for malaria parasite detection in a malaria endemic area | 1 year based on frozen specimens
  based on microscopy of a blood smear or PCR in case of a negative smear or incongruent results. Diagnostic performance will be evaluated before and after training of the algorithm.
  Malaria parasitemia is defined as the presence of one or more parasites in malaria microscopy or a malaria qPCR 18S result over 50 p/ml.
• Diagnostic sensitivity and specificity of Sysmex XN infection manager for diagnosing bacterial bloodstream infection (bBSI) and mixed malaria/bBSI in a malaria endemic area in participants of 5 years and older | 1 year based on frozen specimens
  Diagnostic performance will be evaluated before and after training of the algorithm.
  Malaria parasitemia is defined as the presence of one or more parasites in malaria microscopy or a malaria qPCR 18S result over 50 p/ml Bacterial bloodstream infection is defined as growth of a clinically significant bacterial organism from blood culture within 5 days of incubation or a (16s) PCR result positive for a clinically significant organism.

SECONDARY OUTCOMES:
• Diagnostic performance of the Sysmex XN analyser to diagnose malaria compared to malaria rapid diagnostic test | 1 year based on frozen specimens
  Malaria parasitemia is defined as the presence of one or more parasites in malaria microscopy or a malaria qPCR 18S result over 50 p/ml
• Diagnostic sensitivity and specificity of Sysmex XN analyser to diagnose viral infections or non-bacteremic bacterial infections with or without malaria | 1 year based on frozen specimens
  In participants of 5 years and older. Performance will be tested before and after training the algorithm.
  For description of case definitions, please see detailed description
• Comparison of diagnostic performance of Sysmex XN analyser compared with C-reactive protein and procalcitonin in diagnosing malaria with or without co-infections, bacterial and viral infections. | 1 year based on frozen specimens
  Performance will be tested before and after training the algorithm. For description of case definitions, please see detailed description
• To develop and optimize an algorithm to diagnose viral and bacterial infection in children below 5 years of age. | 1 year based on frozen specimens
  The data will be used to train an algorithm. For description of case definitions, please see detailed description

CONTACTS AND LOCATIONS:
Overall Officials: Andre van der Ven, Principal Investigator — Radboud University Medical Center; Halidou Tinto, Principal Investigator — CRUN; Jan Jacobs, Principal Investigator — ITG
Locations (1):
- Clinical Research Unit Nanaro, Nanaro, Nanaro, Burkina Faso

REFERENCES:
- [Derived] Valia D, Ingelbeen B, Kabore B, Karama I, Peeters M, Lompo P, Vlieghe E, Post A, Cox J, de Mast Q, Robert A, van der Sande MAB, Villalobos HR, van der Ven A, Tinto H, Jacobs J. Use of WATCH antibiotics prior to presentation to the hospital in rural Burkina Faso. Antimicrob Resist Infect Control. 2022 Apr 13;11(1):59. doi: 10.1186/s13756-022-01098-8. PMID 35418154
- [Derived] Post A, Kabore B, Bognini J, Diallo S, Lompo P, Kam B, Herssens N, van Opzeeland F, van der Gaast-de Jongh CE, Langereis JD, de Jonge MI, Rahamat-Langendoen J, Bousema T, Wertheim H, Sauerwein RW, Tinto H, Jacobs J, de Mast Q, van der Ven AJ. Infection Manager System (IMS) as a new hemocytometry-based bacteremia detection tool: A diagnostic accuracy study in a malaria-endemic area of Burkina Faso. PLoS Negl Trop Dis. 2021 Mar 1;15(3):e0009187. doi: 10.1371/journal.pntd.0009187. eCollection 2021 Mar. PMID 33647009
- [Derived] Kabore B, Post A, Berendsen MLT, Diallo S, Lompo P, Derra K, Rouamba E, Jacobs J, Tinto H, de Mast Q, van der Ven AJ. Red blood cell homeostasis in children and adults with and without asymptomatic malaria infection in Burkina Faso. PLoS One. 2020 Nov 30;15(11):e0242507. doi: 10.1371/journal.pone.0242507. eCollection 2020. PMID 33253198
- [Derived] Post A, Kabore B, Reuling IJ, Bognini J, van der Heijden W, Diallo S, Lompo P, Kam B, Herssens N, Lanke K, Bousema T, Sauerwein RW, Tinto H, Jacobs J, de Mast Q, van der Ven AJ. The XN-30 hematology analyzer for rapid sensitive detection of malaria: a diagnostic accuracy study. BMC Med. 2019 May 31;17(1):103. doi: 10.1186/s12916-019-1334-5. PMID 31146732